CLINICAL TRIAL: NCT00423527
Title: Double-blind, Randomised,Placebo-controlled Trial of Levetiracetam in Central Pain in Multiple Sclerosis
Brief Title: Levetiracetam in Central Pain in Multiple Sclerosis(MS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Professor Søren H. Sindrup, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: keppra3
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2007-01

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; central pain; levetiracetam
MeSH Terms: conditions — Multiple Sclerosis | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: levetiracetam — Levetiracetam tablets 500 mg, total daily dose 3000 mg

SUMMARY:
Multiple sclerosis is often associated with pain. There is no standard treatment of this type of pain. Levetiracetam is a new anticonvulsant and it is the hypothesis that it could relieve central pain in multiple sclerosis. This is a randomised, double-blind, placebo-controlled, cross-over trial on the effect of levetiracetam 3000 mg daily on pain in multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* ms diagnosis verified
* age > 18 years
* central pain symptoms for more than 3 months
* central pain diagnosis confirmed by neurological examination
* adequate anticonceptive treatment for women with child bearing potential
* informed consent
* baseline pain of more than 4 on numeric rating scale

Exclusion Criteria:

* other cause of pain
* previous allergic reaction towards levetiracetam
* known adverse drug reaction on levetiracetam
* pregnancy
* severe disease
* inability to follow study protocol
* treatment with antidepressants, other anticonvulsants or opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Pain relief rated on a 0 to 10 point numeric rating scale (median value for last treatment week of each period) | Weekly

SECONDARY OUTCOMES:
Pain rated on a 0 to 10 point numeric rating scale | Daily
Pain subtypes rated on the same scale. | Daily
Brush-evoked pain | Baseline and end of each treatment period
Pin-prick-evoked pain | Daily
Cold-evoked pain | Daily
Health related quality of life (SF36) | Baseline and end of each treatment period
Pain related sleep disturbance | Daily
Use of escape medication | Daily
Muscle spasms as measured on 2 different scales | Baseline and end of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Søren H Sindrup, MD, Principal Investigator — Department of Neurology, Odense Unviersity Hospital
Locations (1):
- Department of Neurology, Odense University Hospital, Odense C, Denmark